CLINICAL TRIAL: NCT01300156
Title: A Multicenter Phase II Study of Etoposide, Methylprednisolone, High-dose Cytarabine and Oxaliplatin (ESHAOx) for Patients With Refractory or Relapsed Hodgkin's Lymphoma (HL)
Brief Title: Etoposide, Methylprednisolone, High-dose Cytarabine and Oxaliplatin (ESHAOx) for Refractory or Relapsed Hodgkin's Lymphoma (HL)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Asan Medical Center (Other); Severance Hospital (Other)
Responsible Party: Hyeon-Seok Eom / MD, PhD, Natioinal Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-10-524
Record Dates: First submitted 2011-02-18; First posted 2011-02-21 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-02

CONDITIONS: Hodgkin's Lymphoma
Keywords: Hodgkin's disease; lymphoma; Relapsed; refractory
MeSH Terms: conditions — Hodgkin Disease; Lymphoma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ESHAOx arm (Experimental): Patients who are planned to be treated with ESHAOx chemotherapy
  Interventions: Drug: Oxaliplatin-based chemotherapy (ESHAOx)

INTERVENTIONS:
Drug: Oxaliplatin-based chemotherapy (ESHAOx) — * Etoposide 40 mg/m2, D1-4
  * Methylprednisolone 500mg, D1-5
  * Cytarabine 2 g/m2, D5
  * Oxaliplatin 130 mg/m2, D1

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of combination chemotherapy with etoposide, methylprednisolone, high-dose cytarabine and oxaliplatin (ESHAOx) for patients with refractory or relapsed Hodgkin's lymphoma (HL).

ELIGIBILITY:
Inclusion Criteria:

* Previously histologically confirmed Hodgkin's lymphoma
* Failure to achieve a complete remission with the initial induction chemotherapy, or recurrent disease
* Performance status (ECOG) ≤ 3
* Age ≤ 75 years old
* Number of prior chemotherapies: one or two regimens
* At least one or more uni-dimensionally measurable lesion(s) defined as; ≥ 2 cm by conventional CT or ≥ 1 cm by spiral CT or skin lesion (photographs should be taken) or measurable lesion by physical examination
* Adequate organ functions defined as; ANC > 1,500/ul, platelet > 75,000/ul, transaminases < 3 X upper normal values; bilirubin < 2 mg/dL
* Written informed consent approved by institutional review board or ethic committee

Exclusion Criteria:

* Previous high dose chemotherapy with autologous stem cell transplantation or allogeneic stem cell transplantation
* Previous chemotherapies with ESHAP regimen
* Any other malignancies within the past 5 years except skin basal cell carcinoma or carcinoma in situ of cervix
* Other serious illness or medical conditions
* Unstable cardiac disease despite treatment, myocardial infarction within 6 months prior to study entry
* History of significant neurologic or psychiatric disorders including dementia or seizures
* Active uncontrolled infection (viral, bacterial or fungal infection)
* Other serious medical illnesses
* Pregnancy or breast-feeding, women of childbearing potential not employing adequate contraception
* Previous history of drug allergy to one of the drugs in the study regimen

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2011-02; Primary Completion 2013-06 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response rate to ESHAOx chemotherapy | within 3 weeks after the completion of the treatment
  To evaluate response rate by Cheson criteria for malignant lymphoma after 3 and 6 cycles of treatment with ESHAOx regimen in patients with refractory or relapsed Hodgkin's lymphoma.

SECONDARY OUTCOMES:
Overall survival, response duration, toxicity profiles | up to 5 years after the completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hyeon Seok Eom, MD, PhD, Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Korea, Goyang, South Korea

REFERENCES:
- [Derived] Won YW, Lee H, Eom HS, Kim JS, Suh C, Yoon DH, Hong JY, Kang HJ, Lee JH, Kim WS, Kim SJ, Lee WS, Chang MH, Do YR, Yi JH, Kim I, Won JH, Kim K, Oh SY, Jo JC. A phase II study of etoposide, methylprednisolone, high-dose cytarabine, and oxaliplatin (ESHAOx) for patients with refractory or relapsed Hodgkin's lymphoma. Ann Hematol. 2020 Feb;99(2):255-264. doi: 10.1007/s00277-019-03891-9. Epub 2020 Jan 2. PMID 31897676